CLINICAL TRIAL: NCT01086085
Title: A Study on Optimizing the Treatment in HBeAg Positive CHB Patients With Response Guide Treatment (RGT) Method.
Brief Title: A Study of Peginterferon Alfa-2a [PEGASYS] in Patients With Chronic Hepatitis B Who Are HBeAg Positive
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Major Science and Technology Special Project of China Eleventh Five-year (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML22266
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — adefovir; peginterferon alfa-2a

ARMS (4):
- A (Experimental)
  Interventions: Drug: peginterferon alfa-2a [PEGASYS]
- B (Experimental)
  Interventions: Drug: peginterferon alfa-2a [PEGASYS]
- C (Experimental)
  Interventions: Drug: peginterferon alfa-2a [PEGASYS]
- D (Experimental)
  Interventions: Drug: Adefovir; Drug: peginterferon alfa-2a [PEGASYS]

INTERVENTIONS:
Drug: Adefovir — Adefovir 10 mg po once daily for 36 weeks
  Arms: D
Drug: peginterferon alfa-2a [PEGASYS] — Early responders: PEGASYS 180 mcg sc once weekly for 48 weeks
  Arms: A
Drug: peginterferon alfa-2a [PEGASYS] — Non-early responders: PEGASYS 180 mcg sc once weekly for 48 weeks
  Arms: B
Drug: peginterferon alfa-2a [PEGASYS] — Non-early responders: PEGASYS 180 mcg sc once weekly for 96 weeks
  Arms: C; D

SUMMARY:
This open-label, multi-center study will evaluate the effect on the quantitative HBsAg reduction of peginterferon alfa-2a [PEGASYS] in patients with HBeAg positive chronic hepatitis B. Patients will receive PEGASYS 180 mcg sc once weekly. After 24 weeks of treatment, rapid responders will receive another 24 weeks of treatment. After 24 weeks of treatment, slow responders will be randomized to another 24 or 72 weeks of PEGASYS monotherapy, or to 72 weeks PEGASYS plus 36 weeks adefovir (10 mg, po once daily, starting from week 29 of PEGASYS treatment). The anticipated time on study drug is >2 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >/=18 years of age
* HBeAg positive chronic hepatitis B
* Compensated liver disease

Exclusion Criteria:

* Patients who had previously received treatment of drugs with activity against HBV within 6 months prior to study start
* Antiviral, anti-neoplastic or immunomodulatory treatment
* Co-infection with active hepatitis A, hepatitis C, hepatitis D, or HIV
* Evidence of decompensated liver disease
* Chronic liver disease other than viral hepatitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2010-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Efficacy: Quantitative HBsAG reduction (proportion of patients with HBsAG reduction) | Weeks 72, 96, 120

SECONDARY OUTCOMES:
Proportion of patients achieving HBeAG seroconversion and HBV DNA </=100000 copies/ml | Weeks 24, 48, 72, 96, 120
Safety: Adverse Events | From baseline to Week 120

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- China (6):
  - Beijing
  - Changchun
  - Guangzhou
  - Shanghai
  - Wuhan
  - Xi'an

REFERENCES:
- [Derived] Sun J, Ma H, Xie Q, Xie Y, Sun Y, Wang H, Shi G, Wan M, Niu J, Ning Q, Yu Y, Zhou H, Cheng J, Kang W, Xie Y, Fan R, Wei L, Zhuang H, Jia J, Hou J. Response-guided peginterferon therapy in patients with HBeAg-positive chronic hepatitis B: A randomized controlled study. J Hepatol. 2016 Oct;65(4):674-682. doi: 10.1016/j.jhep.2016.05.024. Epub 2016 May 26. PMID 27238752